CLINICAL TRIAL: NCT00483236
Title: Quality of Life Measures After Mitral Valve Repair in Non-Ischaemic Cardiomyopathy
Brief Title: Prospective Study Looking at Quality of Life Measures in Non-ischaemic Cardiomyopathy After Mitral Valve Repair
Status: Withdrawn | Type: Observational
Why Stopped: Lack of patient recruitment.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nadia Giannetti, Chief of Cardiology, McGill University Health Center, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: BMB-06-022
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Mitral Valve Insufficiency; Dilated Cardiomyopathy; Congestive Heart Failure
Keywords: Non-Ischaemic Cardiomyopathy
MeSH Terms: conditions — Mitral Valve Insufficiency; Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* Chronic severe mitral regurgitation can lead to symptoms and left ventricular dysfunction.
* The purpose of this study is to prospectively follow patients with non-ischaemic cardiomyopathy who are eligible for mitral valve repair surgery and primarily measure the quality of life through the Minnesota Living with Heart Failure Questionnaire & the Kansas City Cardiomyopathy Questionnaire.

DETAILED DESCRIPTION:
* Chronic mitral regurgitation (MR) usually spirals into a vicious cycle of left ventricular (LV) volume overload, LV dilatation, mitral annular dilatation and more MR. "MR begets MR". Eventually symptoms and LV dysfunction ensue. However, it can often be treated medically or surgically. Medical therapy is primarily afterload reduction and diuretics. Surgically, there are two options, either mitral valve repair or replacement.
* A number of retrospective studies have demonstrated improved LV function and survival in patients undergoing valve repair compared to valve replacement with or without subvalvular preservation. In one report, for example, patients who underwent valve repair were compared to patients who underwent valve replacement. The report found that the former group had lower operative mortality, a greater increase in LV ejection fraction and higher overall ten year survival.
* The bulk of the literature at present addresses left ventricular dimensions, ejection fraction, geometry and New York Heart Association functional class, but few have addressed quality of life measures. In addition, most of these studies were retrospective and the majority of patients had concomitant ischaemic heart disease.
* Even though the studies concerning quality of life after mitral valve surgery have been few, nevertheless, some have addressed isolated valve surgery without concomitant bypass surgery and have shown improved quality of life, though follow up in some was limited to 3 months. We will follow our population for 12 months after surgical repair.
* We will primarily look at subjective measures for quality of life such as the Minnesota Living with Heart Failure Questionnaire & the Kansas City Cardiomyopathy Questionnaire, as subjective measures are becoming more and more important following cardiac surgery. Patients will serve as their own controls and all study parameters will be compared pre- and post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that fulfill surgical criteria set by the 2006 ACC/AHA guidelines for the management of patients with valvular heart disease.
* Symptomatic mitral regurgitation with left ventricular dysfunction (LVEF < or = 40%) on maximal medical therapy

Exclusion Criteria:

* Mitral valve replacement
* Concomitant coronary artery bypass surgery
* Patient unable to give informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart Failure Clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-12-01 (Estimated); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life scores as measured by the Minnesota Living with Heart Failure Questionnaire & the Kansas City Cardiomyopathy Questionnaire | 12 months

SECONDARY OUTCOMES:
1- Echocardiographic parameters 2- 6 minute walk test 3- NYHA class 4- Hospitalisation for heart failure, redo surgery, morbidity & mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Giannetti, MD.,FRCPC, Principal Investigator — Director of Heart Failure and Transplant Centre at McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada